CLINICAL TRIAL: NCT01525069
Title: Pilot Study of Hepatic Arterial Infusion Therapy in Patients With Unresectable or Borderline Resectable Intrahepatic Cholangiocarcinoma
Brief Title: Hepatic Arterial Infusion in Treating Patients With Locally Advanced, Non-Metastatic Cholangiocarcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Equipment that was used in the study was discontinued
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201111068
Record Dates: First submitted 2012-01-25; First posted 2012-02-02 (Estimated); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Cholangiocarcinoma; Liver Neoplasms
MeSH Terms: conditions — Cholangiocarcinoma; Liver Neoplasms | interventions — Floxuridine; Dexamethasone; Calcium Dobesilate; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A (HAI FUDR alone) (Experimental): * 14-42 days after surgery for insertion of the HAI pump, floxuridine (FUDR) and dexamethasone plus heparin in normal saline to a total volume of 30 ml will be administered through the HAI pump.
  * This will be repeated on Day 1 of each 28 day cycle. FUDR administration will be a 14-day continuous infusion using the HAI pump.
  * The pump will be emptied and refilled with heparinized normal saline and dexamethasone on Day 15 of each cycle to be infused over the next 14 days.
  Interventions: Drug: Floxuridine; Drug: Dexamethasone
- Arm B (HAI FUDR + gemcitabine) (Experimental): * Consists of Cohort B1, B2, and B3. Enrollment to specific cohorts will depend on the number of DLTs in each cohort. Each cohort has a different dose of FUDR and gemcitabine.
  * Gemcitabine IV will be given on Days 1, 8, and 15 of each 28 day cycle in Cohort B1
  * Gemcitabine IV will be given on Days 1 and 15 of each 28 day cycle in Cohort B2 & B3
  * 14-42 days after surgery for insertion of the HAI pump, floxuridine (FUDR) and dexamethasone plus heparin in normal saline to a total volume of 30 ml will be administered through the HAI pump.
  * This will be repeated on Day 1 of each 28 day cycle. FUDR administration will be a 14-day continuous infusion using the HAI pump.
  * The pump will be emptied and refilled with heparinized normal saline and dexamethasone on Day 15 of each cycle to be infused over the next 14 days.
  Interventions: Drug: Floxuridine; Drug: Dexamethasone; Drug: Gemcitabine
- Arm C (HAI FUDR + gemcitabine + oxaliplatin) (Experimental): * Consists of Cohort C1, C2, C3, and C4. Enrollment to specific cohorts will depend on the number of DLTs in each cohort. Each cohort has a different dose of FUDR, gemcitabine, and oxaliplatin.
  * Gemcitabine IV will be given on Days 1 and 15 of each 28 day cycle.
  * Oxaliplatin IV will be given on Days 1 and 15 of each 28 days cycle.
  * 14-42 days after surgery for insertion of the HAI pump, floxuridine (FUDR) and dexamethasone plus heparin in normal saline to a total volume of 30 ml will be administered through the HAI pump.
  * This will be repeated on Day 1 of each 28 day cycle. FUDR administration will be a 14-day continuous infusion using the HAI pump.
  * The pump will be emptied and refilled with heparinized normal saline and dexamethasone on Day 15 of each cycle to be infused over the next 14 days.
  Interventions: Drug: Floxuridine; Drug: Dexamethasone; Drug: Gemcitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Floxuridine
  Other Names: 5-FUDR, FdUrD, floxuridin, fluorodeoxyuridine, fluoruridine deoxyribose, FUdR
Drug: Dexamethasone
  Other Names: Aeroseb-Dex, Decaderm, Decadron, Decaspray, DM, DXM
Drug: Gemcitabine
  Other Names: dFdC, dFdCyd, difluorodeoxycytidine hydrochloride, gemcitabine, Gemzar, LY-188011
  Arms: Arm B (HAI FUDR + gemcitabine); Arm C (HAI FUDR + gemcitabine + oxaliplatin)
Drug: Oxaliplatin
  Other Names: 1-OHP, Dacotin, Dacplat, diaminocyclohexane oxalatoplatinum, Eloxatin, L-OHP
  Arms: Arm C (HAI FUDR + gemcitabine + oxaliplatin)

SUMMARY:
This pilot clinical trial studies the safety and effectiveness of continuous hepatic arterial infusion (HAI) of floxuridine (FUDR) alone or in combination with other chemotherapeutic drugs in treating patients with locally advanced cholangiocarcinoma that cannot be removed by surgery. HAI is a method to deliver higher concentrations of FUDR more directly to liver tumors and reduces side effects. HAI alone or in combination with oxaliplatin and/or gemcitabine may significantly improve clinical outcomes of patients with locally advanced cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have suspected intrahepatic or hilar cholangiocarcinoma with minimal extrahepatic disease. Diagnosis must be histologically or cytologically confirmed for continued treatment on study after pump placement.
* Patient must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan/MRI
* Patient must have disease that is unresectable or borderline resectable with < 70% liver involvement by cancer
* Patient must be >= 18 years old.
* Patient's Eastern Cooperative Oncology Group (ECOG) performance status must be =< 2 (Karnofsky >= 60%)
* Patient must have normal organ and marrow function as defined below:

  * Absolute neutrophil count >= 1,500/mcL
  * Platelets >= 75,000/mcL
  * Total bilirubin =< 2 mg/dL
  * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 5 X institutional upper limit of normal
  * Creatinine <= institutional upper limit normal
* Patient must be able to understand and willing to sign a written informed consent document

Exclusion Criteria:

* Patients must not have had prior treatment with FUDR
* Patient must not be receiving any other investigational agents
* Patient must not have a diagnosis of Gilbert's disease
* Patient must not have a diagnosis of hepatic encephalopathy
* Patient must not have had prior external beam radiation to the liver
* Patient must not have a diagnosis of sclerosing cholangitis
* Patient must not have any uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patient must not be pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-04-03 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) | Completion of 2 cycles of treatment by all patients (approximately 4 years)
  Document the frequency of grades 3-5 non-hematologic toxicities (dose-limiting toxicities) associated with the treatment regimen by patient and by type of toxicity for each cohort during the first 2 cycles of treatment

SECONDARY OUTCOMES:
Time to progression (TTP) | 12 months
  Describe median time to progression with a 95% confidence interval for each cohort.
Response rates | 8 weeks
  The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started)
  Using RECIST 1.1
Overall survival | 12 months
Number and grade of adverse events | Beginning with pump placement and continuing for 30 days following the last day of study treatment (median length of treatment 3 months)
  Determine safety, tolerability and toxicities based on the number and grade of adverse events associated with this regimen.
Imaging biomarkers of tumor response | Pre-treatment and then every 8 weeks during treatment (median length of treatment 3 months)
  Using magnetic resonance diffusion-weighted imaging (DW-MRI) and dynamic contrast enhanced magnetic resonance imaging (DCE-MRI) before and during the course of treatment with HAI therapy, validate imaging biomarkers of tumor response
Overall survival | Up to 5 years
Time to progression (TTP) | 24 months
  Describe median time to progression with a 95% confidence interval for each cohort.

CONTACTS AND LOCATIONS:
Overall Officials: William Chapman, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valle JW WH, Palmer DD, Cunningham D, Anthoney DA, Maraveyas A, Hughes SK, Roughton JA, Bridgewater JA: Gemcitabine with or without cisplatin in patients (pts) with advanced or metastatic biliary tract cancer (ABC): Results of a multicenter, randomized phase III trial (the UK ABC-02 trial). J Clin Oncol 27:15s, 2009 (suppl, abstr 4503), 2009
- [Background] Tan BR, Brenner WS, Picus J, Marsh S, Gao F, Fournier C, Fracasso PM, James J, Yen-Revollo JL, McLeod HL. Phase I study of biweekly oxaliplatin, gemcitabine and capecitabine in patients with advanced upper gastrointestinal malignancies. Ann Oncol. 2008 Oct;19(10):1742-8. doi: 10.1093/annonc/mdn375. Epub 2008 Jun 4. PMID 18534963
- [Background] Kemeny NE, Melendez FD, Capanu M, Paty PB, Fong Y, Schwartz LH, Jarnagin WR, Patel D, D'Angelica M. Conversion to resectability using hepatic artery infusion plus systemic chemotherapy for the treatment of unresectable liver metastases from colorectal carcinoma. J Clin Oncol. 2009 Jul 20;27(21):3465-71. doi: 10.1200/JCO.2008.20.1301. Epub 2009 May 26. PMID 19470932
- [Background] Kemeny NE, Gonen M. Hepatic arterial infusion after liver resection. N Engl J Med. 2005 Feb 17;352(7):734-5. doi: 10.1056/NEJM200502173520723. No abstract available. PMID 15716576
- [Background] Jarnagin WR, Schwartz LH, Gultekin DH, Gonen M, Haviland D, Shia J, D'Angelica M, Fong Y, DeMatteo R, Tse A, Blumgart LH, Kemeny N. Regional chemotherapy for unresectable primary liver cancer: results of a phase II clinical trial and assessment of DCE-MRI as a biomarker of survival. Ann Oncol. 2009 Sep;20(9):1589-1595. doi: 10.1093/annonc/mdp029. Epub 2009 Jun 2. PMID 19491285
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu